CLINICAL TRIAL: NCT01405092
Title: Continuous Versus Conventional Volume Management During CRRT (Continuous Renal Replacement Therapy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Devasmita C. Dev MD, Director of In-center and Home Dialysis, Dallas VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: #09-097
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Continuous Renal Replacement Therapy
Keywords: volume; acute kidney injury; continuous renal replacement
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard volume management (Placebo Comparator): patients on this arm will receive usual care volume management during continuous renal replacement therapy
  Interventions: Device: use of continuous renal replacement machine for renal replacement
- continuous volume management (Active Comparator): use of Critline, Hemametrics USA, in conjunction with continuous renal replacment therapy to determine volume removal
  Interventions: Device: use of continuous renal replacement machine for renal replacement; Device: use of blood volume monitoring device in conjunction with machine used for continuous renal replacement to assess and determine volume removal

INTERVENTIONS:
Device: use of continuous renal replacement machine for renal replacement — usual care with volume removal during continuous renal replacement therapy
Device: use of blood volume monitoring device in conjunction with machine used for continuous renal replacement to assess and determine volume removal — blood volume monitoring device, Critline, Hemametric, USA, will be used in conjunction with continuous renal replacement to determine rate of volume removal
  Arms: continuous volume management

SUMMARY:
Use of on-line blood volume monitoring during continuous renal replacement therapy can improve volume management in acute kidney injury patients requiring renal replacement

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney injury requiring continuous renal replacement therapy and volume removal

Exclusion Criteria:

* unable to provide or obtain patient consent
* not expected to survive 48 hours

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
compare number of hypotensive events in treatment versus control arms | 24 hour for each arm
  compare the number of hypotensive events during use of crit-line monitor over 24 hour period versus during control 24 hour period

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States